CLINICAL TRIAL: NCT03095066
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Neurobehavioral Disinhibition Including Aggression, Agitation, and Irritability in Patients With Traumatic Brain Injury (TBI).
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Neurobehavioral Disinhibition Including Aggression, Agitation, and Irritability in Participants With Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-AVP-786-205
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Neurobehavioral Disinhibition
Keywords: aggression; agitation; irritability; non-penetrating brain injury; traumatic brain injury; TBI; AVP-786
MeSH Terms: conditions — Aggression; Psychomotor Agitation; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Overall Study: Stage 1 Placebo/Stage 2 Placebo or Stage 1 Placebo/Stage 2 AVP-786 (Placebo Comparator): Participants received AVP-786 matching placebo capsules, orally, twice daily (BID) during Weeks 1 to 6 of the Stage 1 treatment period. After Week 6 participants were classified as responders or non-responders and were re-randomized to receive either placebo, orally, BID or AVP-786 in a dose escalation schedule to reach the target dose of AVP-786-42.63/4.9, orally, BID during Week 7 to Week 12 of Stage 1 treatment period.
  Interventions: Drug: Placebo; Drug: AVP-786-42.63
- Overall Study: Stage 1 AVP-786/Stage 2 AVP-786 (Experimental): Participants received AVP-786-28/4.9 (deudextromethorphan hydrobromide (d6-DM) 28 milligrams (mg)/quinidine sulfate (Q) 4.9 mg) capsule, along with AVP-786 matching placebo capsule, orally, once daily (QD) during Week 1 followed by AVP-786-28/4.9 capsule, orally, BID during Week 2, and AVP-786-42.63/4.9 (d6-DM 42.63 mg/Q 4.9 mg) capsules (target dose), orally, BID during Weeks 3 to 12 of the treatment period.
  Interventions: Drug: Placebo; Drug: AVP-786-28; Drug: AVP-786-42.63
- Stage 1: Placebo (Placebo Comparator): Participants received AVP-786 matching placebo capsules, orally, BID during Weeks 1 to 6 of the Stage 1 treatment period.
  Interventions: Drug: Placebo
- Stage 1: Placebo Non-responders to Stage 2: Placebo (Placebo Comparator): Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders (responders" if modified Clinical Global Impression of Severity [mCGI-S] score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week 6 were re-randomized to continue receiving AVP-786 matching placebo capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
  Interventions: Drug: Placebo
- Stage 1: Placebo Non-responders to Stage 2: AVP-786 (Experimental): Participants who received placebo in Stage 1 and were classified as non-responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week 6 were re-randomized to receive AVP-786 in Stage 2 using the same dose escalation schedule used in Stage 1 i.e., AVP-786-28- 28/4.9 capsule, along with AVP-786 matching placebo capsule, orally, QD during Week 7 followed by AVP-786-28 -28/4.9 capsule, orally, BID during Week 8, and AVP-786-42.63/4.9 capsules, orally, BID during Weeks 9 to 12 of the Stage 2 treatment period.
  Interventions: Drug: Placebo; Drug: AVP-786-28; Drug: AVP-786-42.63
- Stage 1: Placebo Responders to Stage 2: Placebo (Placebo Comparator): Participants who were randomized to receive placebo in Stage 1 and were classified as responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline) after Week 6 were re-randomized to continue receiving AVP-786 matching placebo capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
  Interventions: Drug: Placebo
- Stage 1: Placebo Responders to Stage 2: AVP-786 (Experimental): Participants who received placebo in Stage 1 and were classified as responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline) after Week 6 were re-randomized to receive AVP-786 in Stage 2 using the same dose escalation schedule used in Stage 1 i.e., AVP-786-28- 28/4.9 capsule, along with AVP-786 matching placebo capsule, orally, QD during Week 7 followed by AVP-786-28 -28/4.9 capsule, orally, BID during Week 8, and AVP-786-42.63/4.9 capsules, orally, BID during Weeks 9 to 12 of the Stage 2 treatment period.
  Interventions: Drug: Placebo; Drug: AVP-786-28; Drug: AVP-786-42.63
- Stage 1: AVP-786 (Experimental): Participants received AVP-786-28/4.9 (deudextromethorphan hydrobromide (d6-DM) 28 milligrams (mg)/quinidine sulfate (Q) 4.9 mg) capsule, along with AVP-786 matching placebo capsule, orally, once daily (QD) during Week 1 followed by AVP-786-28/4.9 capsule, orally, BID during Week 2, and AVP-786-42.63/4.9 (d6-DM 42.63 mg/Q 4.9 mg) capsules (target dose), orally, BID during Weeks 3 to 6 of the Stage 1 treatment period.
  Interventions: Drug: Placebo; Drug: AVP-786-28; Drug: AVP-786-42.63

INTERVENTIONS:
Drug: Placebo — Administered as capsules
Drug: AVP-786-28 — 28 mg of d6-DM and 4.9 mg of Q
  Arms: Overall Study: Stage 1 AVP-786/Stage 2 AVP-786; Stage 1: AVP-786; Stage 1: Placebo Non-responders to Stage 2: AVP-786; Stage 1: Placebo Responders to Stage 2: AVP-786
Drug: AVP-786-42.63 — 42.63 mg of d6-DM and 4.9 mg of Q
  Arms: Overall Study: Stage 1 AVP-786/Stage 2 AVP-786; Overall Study: Stage 1 Placebo/Stage 2 Placebo or Stage 1 Placebo/Stage 2 AVP-786; Stage 1: AVP-786; Stage 1: Placebo Non-responders to Stage 2: AVP-786; Stage 1: Placebo Responders to Stage 2: AVP-786

SUMMARY:
This is a multicenter, randomized, placebo-controlled study to evaluate AVP-786 for the treatment of neurobehavioral disinhibition including aggression, agitation, and irritability in participants with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Eligible participants for this study must have a diagnosis of neurobehavioral disinhibition including aggression, agitation, and irritability that persists after brain injury.

This is a multicenter, randomized, placebo-controlled study, consisting of up to 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with TBI
* Participants with neurobehavioral disinhibition symptoms that are present after trauma or after recovery of consciousness
* Score of ≥4 on the mCGI-S scale and the Agitation/Aggression or Irritability/Lability subscales of the Neuropsychiatric Inventory (NPI) scale at screening and baseline
* Participants with a reliable caregiver

Exclusion Criteria:

* Participants with significant symptoms of a major depressive disorder
* Participants with a history of or current clinical symptoms of schizophrenia, schizoaffective disorder, bipolar disorder, antisocial personality disorder, or borderline personality disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Tuscaloosa Veterans Affairs Medical Center, Tuscaloosa, Alabama
  - Absolute Clinical Research Site#207, Phoenix, Arizona
  - Perseverance Research Center Site#152, Scottsdale, Arizona
  - ATP Clinical Research Site#150, Costa Mesa, California
  - Kaizen Brain Center #224, La Jolla, California
  - Sunwise Clinical Research, LLC Site#216, Lafayette, California
  - Torrance Clinical Research Institute Site#157, Lomita, California
  - Tibor Rubin VA Medical Center, SCIRE Biomedical Research Institute, Long Beach, California
  - Asclepes Research Centers - Panorama City Site #208, Panorama City, California
  - The Neurology Group, Pomona, California
  - Mountain Mind, Colorado Springs, Colorado
  - Mountain View Clinical Research, Inc. Site# 202, Denver, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Bradenton Research Center, Inc, Bradenton, Florida
  - Healthcare Innovative Institute, LLC Site# 173, Coral Springs, Florida
  - Science Connections, LLC Site#161, Doral, Florida
  - Design Neuroscience Center, PL, Doral, Florida
  - Alphab Global Research Site#163, Jupiter, Florida
  - Meridien Research, Maitland, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Project 4 Research, Miami, Florida
  - Allied Biomedical Research Institute, Inc. Site#151, Miami, Florida
  - Health Synergy Clinical Research, Okeechobee, Florida
  - Roskamp Institute Clinic, Inc., Sarasota, Florida
  - USF Dept of Psychiatry and Behavioral Neurosciences Site# 214, Tampa, Florida
  - Meridien Research Site# 108, Tampa, Florida
  - Hawaii Pacific Neuroscience Site#184, Honolulu, Hawaii
  - The University of Kentucky research foundation, Lexington, Kentucky
  - Baptist Health, Richmond, Kentucky
  - Sisu BHR Site#200, Springfield, Massachusetts
  - Neurobehavioral Medicine Group #222, Bloomfield Hills, Michigan
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Sharlin Health and Neurology, Ozark, Missouri
  - Clinical Research Professionals, St Louis, Missouri
  - JFK Johnson Rehabilitation Institute, Edison, New Jersey
  - The NeuroCognitive Insititute, Mount Arlington, New Jersey
  - New York University School of Medicine Site #122, New York, New York
  - Atrium Health - Carolinas Rehabilitation - Charlotte Site #166, Charlotte, North Carolina
  - New Hope Clinical Research Site#194, Charlotte, North Carolina
  - Carolina Headache Institute, Durham, North Carolina
  - Salisbury VAMC, Salisbury, North Carolina
  - Valley Medical Research, Centerville, Ohio
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - North Star Medical Research, LLC Site#154, Middleburg Heights, Ohio
  - IPS Research Site#196, Oklahoma City, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - WJB Dorn VA-Wm. Jennings Bryan Dorn VA Medical Center, Columbia, South Carolina
  - University of Texas Southwestern Medical Site#140, Dallas, Texas
  - Polytrauma Rehabilitation Center S. Texas VA Health Care System Site# 146, San Antonio, Texas
  - Cedar Clinical Research #221, Draper, Utah
  - Virginia Commonwealth University #172, Richmond, Virginia
  - Virginia Commonwealth University Site#172, Richmond, Virginia
  - Salem Research Institute Site# 138, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 67 investigative sites in the United States from 30 May 2017 to 31 August 2022. A total of 467 participants were screened of which 168 participants were randomized to receive placebo or AVP-786.
Pre-assignment Details: Study was conducted in 2 Stages. Participants randomized to receive placebo in Stage 1 were re-randomized after Week 6 to receive either placebo or AVP-786 in Stage 2. As pre-specified in protocol, participants randomized to 'AVP-786' arm were not re-randomized after Week 6 and continued receiving AVP-786 in the same arm throughout 12 weeks of study. Study is presented in 3 stages: Overall Study, Stage 1 & Stage 2.
Groups:
- Stage 1 and 2: AVP-786: Participants received AVP-786-28/4.9 (deudextromethorphan hydrobromide (d6-DM) 28 milligrams (mg)/quinidine sulfate (Q) 4.9 mg) capsule, along with AVP-786 matching placebo capsule, orally, once daily (QD) during Week 1 followed by AVP-786-28/4.9 capsule, orally, BID during Week 2, and AVP-786-42.63/4.9 (d6-DM 42.63 mg/Q 4.9 mg) capsules (target dose), orally, BID during Weeks 3 to 6 of the Stage 1 treatment period. Participants who completed Stage 1, continued to receive AVP-786-42.63/4.9 (d6-DM 42.63 mg/Q 4.9 mg) capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
Period: Overall Study (Baseline to Week 12)
Arm/Group | Overall Study: Stage 1 Placebo/Stage 2 Placebo or Stage 1 Placebo/Stage 2 AVP-786 | Overall Study: Stage 1 AVP-786/Stage 2 AVP-786 | Stage 1: Placebo | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786 | Stage 1: Placebo Responders to Stage 2: Placebo | Stage 1: Placebo Responders to Stage 2: AVP-786 | Stage 1 and 2: AVP-786
Started (Number 'started' represents participants randomized on Day 1 of the study to receive either AVP-786 or AVP-786 matching placebo.) | 83 | 85 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 58 (Number 'completed' represent the number of participants who completed the entire 12 weeks of the study irrespective of whether they completed the study in Stage 1 or Stage 2.) | 68 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 25 | 17 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Trial Site Terminated by Sponsor | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 8 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 1 (Baseline to Week 6)
Arm/Group | Overall Study: Stage 1 Placebo/Stage 2 Placebo or Stage 1 Placebo/Stage 2 AVP-786 | Overall Study: Stage 1 AVP-786/Stage 2 AVP-786 | Stage 1: Placebo | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786 | Stage 1: Placebo Responders to Stage 2: Placebo | Stage 1: Placebo Responders to Stage 2: AVP-786 | Stage 1 and 2: AVP-786
Started | 0 | 0 | 83 (Number 'started' represent the number of participants who were randomized to receive AVP-786 matching placebo in Stage 1 of the study.) | 0 | 0 | 0 | 0 | 85 (Number 'started' represent the number of participants who were randomized to receive AVP-786 in Stage 1 of the study.)
Completed | 0 | 0 | 68 (Number 'completed' represent the number of participants randomized to receive AVP-786 matching placebo and completed Stage 1 i.e., first 6 weeks of the study.) | 0 | 0 | 0 | 0 | 71
Not Completed | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 14
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance With Study Drug | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Not completed — Trial Site Terminated by Sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Stage 2 (Week 7 to Week 12)
Arm/Group | Overall Study: Stage 1 Placebo/Stage 2 Placebo or Stage 1 Placebo/Stage 2 AVP-786 | Overall Study: Stage 1 AVP-786/Stage 2 AVP-786 | Stage 1: Placebo | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786 | Stage 1: Placebo Responders to Stage 2: Placebo | Stage 1: Placebo Responders to Stage 2: AVP-786 | Stage 1 and 2: AVP-786
Started | 0 | 0 | 0 | 22 (Number 'started' represent the number participants who were classified as 'non-responder' after Week 6 and were re-randomized to continue receiving AVP-786 matching placebo in Stage 2 of the study.) | 17 (Number 'started' represent the number participants who were classified as 'non-responder' after Week 6 and were re-randomized to receive the study drug i.e., AVP-786 in Stage 2 of the study.) | 16 (Number 'started' represent the number participants who were classified as 'responder' after Week 6 and were re-randomized to continue receiving AVP-786 matching placebo in Stage 2 of the study.) | 13 (Number 'started' represent the number participants who were classified as 'responder' after Week 6 and were re-randomized to receive the study drug i.e., AVP-786 in Stage 2 of the study.) | 71 (Number 'started' represent the number of participants who completed Stage 1 and continued to receive the study drug i.e., AVP-786 in Stage 2 of the study.)
Completed (Number 'completed' represent the number of participants who completed Stage 2 i.e., Week 7 to Week 12 of the study.) | 0 | 0 | 0 | 20 | 13 | 14 | 11 | 68
Not Completed | 0 | 0 | 0 | 2 | 4 | 2 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Reason Not Specified | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study medication.
Groups:
- Overall Study: Placebo: Participants received AVP-786 matching placebo capsules, orally, BID during Weeks 1 to 6 of the Stage 1 treatment period. After Week 6 participants were classified as responders or non-responders and were re-randomized to receive either placebo, orally, BID or AVP-786 in a dose escalation schedule to reach the target dose of AVP-786-42.63/4.9, orally, BID during Week 7 to Week 12 of Stage 1 treatment period.
- Overall Study: AVP-786: Participants received AVP-786-28/4.9 (d6-DM 28 mg/ Q 4.9 mg) capsule, along with AVP-786 matching placebo capsule, orally, QD during Week 1 followed by AVP-786-28/4.9 capsule, orally, BID during Week 2, and AVP-786-42.63/4.9 (d6-DM 42.63 mg/Q 4.9 mg) capsules (target dose), orally, BID during Weeks 3 to 12 of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Overall Study: Placebo | Overall Study: AVP-786 | Total
Number analyzed (Participants) | 83 | 85 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.54) | 46.8 (13.93) | 47.1 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 56 | 58 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 79 | 147
  Black or African American | 10 | 3 | 13
  Asian | 2 | 1 | 3
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 27 | 52
  Not Hispanic or Latino | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Change From Baseline in the Composite of the Clinical Impression Severity Scores on the Neuropsychiatric Inventory Clinician Rating Scale (NPI-C) Subscale of Aggression, Agitation, and Irritability/Lability (NPI-C-3)
Description: NPI-C is a retrospective informant/caregiver interview covering 12 neuropsychiatric symptom domains. These are collectively rated first by the informant/caregiver based on frequency (0-4);severity (0-3);informant/caregiver distress (0-5) & then by the participant based on frequency (0-4), which the clinician then integrates into a (0-3) clinical impression severity rating. NPI-C-3= aggression, agitation, & irritability/lability subscales. NPI-C agitation domain= sum of clinical impression severity scores for agitation questions 1-13 (score=0-39). NPI-C aggression domain= sum of clinician impression severity scores for aggression questions 1-8 (score=0-24). NPI-C irritability/lability domain= sum of clinician impression severity scores for irritability/lability questions 1-12 (score=0-36). NPI-C-3 composite score ranges from 0-99. Higher score= increased severity. Least square (LS) mean was analyzed using mixed effects model repeated measures (MMRM) analysis.
Time Frame: Baseline to Week 6
Population: Modified intent-to-treat (mITT) population. Stage 1: Participants randomized in Stage 1 who took at least 1 dose of study medication & had at least 1 post-baseline NPI-C-3 composite score efficacy assessment in Stage 1. Overall number analyzed=participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786
Number analyzed (Participants) | 64 | 61
score on a scale | -18.7 (1.74) | -20.4 (1.73)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Treatment differences in each stage were estimated by the Mixed Model Repeated Measures (MMRM); Test type: Superiority; p = 0.405, MMRM — MMRM included fixed effects of treatment, site, visit, treatment-by-visit interaction, baseline NPI-C-3 value and baseline-by-visit interaction; Difference in LS Mean = -1.7, 95% CI 2-sided [-5.8 to 2.4]

2. Primary Outcome: Stage 2: Change From Baseline in the Composite of the Clinical Impression Severity Scores on the NPI-C Subscale of NPI-C-3
Description: NPI-C is a retrospective informant/caregiver interview covering 12 neuropsychiatric symptom domains. These domains are collectively rated by the informant/caregiver based on frequency (0-4), severity (0-3) & informant/caregiver distress (0-5), then by participant based on frequency (0-4), which is integrated by clinician into (0-3) clinical impression severity rating. NPI-C-3=aggression, agitation, & irritability/lability subscales. NPI-C agitation domain=sum of clinical impression severity scores for agitation questions 1-13 (score=0-39). NPI-C aggression domain=sum of clinician impression severity scores for aggression questions 1-8 (score=0-24). NPI-C irritability/lability domain=sum of clinician impression severity scores for irritability/lability questions 1-12 (score= 0-36). NPI-C-3 composite score ranges from 0-99. Higher score=increased severity. LS mean was analyzed using MMRM analysis. Overall number analyzed=number of participants with data available for analysis.
Time Frame: Week 7 to Week 12
Population: mITT population. Stage 2: participants randomized into Stage 2 with at least 1 NPI-C-3 efficacy assessment in Stage 2. As pre-specified in protocol, data for placebo non-responders re-randomized into Stage 2 was used to estimate & report Stage 2 efficacy. Hence only these Stage 2 arms are reported for the OM.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Stage 1: Placebo Non-responders to Stage 2: Placebo: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score hasdecreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week 6 were re-randomized to continue receiving AVP-786 matching placebo capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
- Stage 1: Placebo Non-responders to Stage 2: AVP-786: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week 6 were re-randomized to receive AVP-786 in Stage 2 using the same dose escalation schedule used in Stage 1 i.e., AVP-786-28/4.9 capsule, along with AVP-786 matching placebo capsule, orally, QD during Week 7 followed by AVP-786-28/4.9 capsule, orally, BID during Week 8, and AVP-786-42.63/4.9 capsules, orally, BID, during Weeks 9 to 12 of the Stage 2 treatment period.
Arm/Group | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 15 | 12
score on a scale | -5.2 (4.97) | -5.9 (5.28)
Statistical Analysis 1: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.921, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = -0.7, 95% CI 2-sided [-15.3 to 13.9]

3. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in NPI-C Rating Scale Subscale Scores for Aggression
Description: The NPI-C was used to rate the presence of neuropsychiatric symptoms across 12 domains. The 12 domains are collectively rated first by the informant/caregiver based on frequency (0-4), severity (0-3) & informant/caregiver distress (0-5), then by the participant based on frequency (0-4), which the clinician then integrates into a (0-3) clinical impression severity rating. The NPI-C aggression domain score is the sum of clinician impression severity scores for aggression questions 1-8, score ranges from 0-24, where higher score indicates greater clinical severity of symptom. LS mean was analyzed using MMRM analysis. Overall number analyzed= number of participants with data available for analysis. Number analyzed= number of participants with data available for analysis at the specified time point.
Time Frame: Stage 1: Baseline to Week 6; Stage 2: Week 7 to Week 12
Population: mITT population. Stage 1:all participants randomized in Stage 1 who took at least 1 dose of study medication &had at least 1 post-baseline NPI-C-3 composite score efficacy assessment in Stage 1; Stage 2:participants randomized into Stage 2 &had at least 1 NPI-C-3 efficacy assessment in Stage 2(after Week 6). As pre-specified in protocol data for placebo non-responders re-randomized into Stage 2 was used to estimate & report Stage 2 efficacy. Hence only these Stage 2 arms are reported for the OM.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Stage 1: Placebo Non-responders; to Stage 2: Placebo: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week 6 were re-randomized to continue receiving AVP-786 matching placebo capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders; to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 64 | 61 | 15 | 12
score on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 64 | 61 | 0 | 0
  Change from Baseline to Week 6 | -3.6 (0.40) | -4.3 (0.40) |  |
  Change from Week 7 to Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Change from Week 7 to Week 12 |  |  | -0.8 (1.39) | -0.6 (1.55)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.150, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = -0.7, 95% CI 2-sided [-1.7 to 0.3]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders; to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.921, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = 0.2, 95% CI 2-sided [-4.3 to 4.7]

4. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in NPI-C Rating Scale Subscale Scores for Agitation
Description: The NPI-C is used to rate the presence of neuropsychiatric symptoms across 12 domains. The 12 domains are collectively rated first by the informant/caregiver based on frequency (0-4), severity (0-3) & informant/caregiver distress (0-5), then by the participant based on frequency (0 to 4), which the clinician then integrates into a (0-3) clinical impression severity rating. The NPI-C agitation domain score is the sum of clinician impression severity scores for agitation questions 1-13, score ranges from 0-39, where higher score indicates greater clinical severity of symptom. LS mean was analyzed using MMRM analysis. Overall number analyzed=number of participants with data available for analysis. Number analyzed=number of participants with data available for analysis at the specified time point.
Time Frame: Stage 1: Baseline to Week 6; Stage 2: Week 7 to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Stage 1: Placebo Non-responders to Stage 2: Placebo: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week 6 were re-randomized to continue receiving AVP-786 matching placebo capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 64 | 61 | 15 | 12
score on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 64 | 61 | 0 | 0
  Change from Baseline to Week 6 | -7.0 (0.69) | -6.7 (0.67) |  |
  Change from Week 7 to Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Change from Week 7 to Week 12 |  |  | -2.6 (1.95) | -0.6 (2.02)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.702, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = 0.3, 95% CI 2-sided [-1.3 to 1.9]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.469, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = 2.0, 95% CI 2-sided [-3.6 to 7.6]

5. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in NPI-C Rating Scale Subscale Scores for Irritability/Lability
Description: NPI-C is used to rate the presence of neuropsychiatric symptoms across 12 domains. The 12 domains are collectively rated first by the informant/caregiver based on frequency (0-4), severity (0-3) & informant/caregiver distress (0-5), then by the participant based on frequency (0 to 4), which the clinician then integrates into a (0-3) clinical impression severity rating. NPI-C irritability/lability domain score=sum of clinician impression severity scores for irritability/lability questions 1-12, score ranges from 0-36, where higher score indicates greater clinical severity of symptom. LS mean was analyzed using MMRM analysis. Overall number analyzed=number of participants with data available for analysis. Number analyzed=number of participants with data available for analysis at the specified time point.
Time Frame: Stage 1: Baseline to Week 6; Stage 2: Week 7 to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Stage 1: Placebo Non-responders to Stage 2: Placebo: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders (responders" if mCGI-S score is ≤ 3 at Day 43 and NPI-C-3 score has decreased by ≥ 25% from baseline. Participants who did not meet these criteria were considered "non-responders) after Week were re-randomized to continue receiving AVP-786 matching placebo capsules, orally, BID during Weeks 7 to 12 of the Stage 2 treatment period.
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 64 | 61 | 15 | 12
score on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 64 | 61 | 0 | 0
  Change from Baseline to Week 6 | -8.5 (0.94) | -9.7 (0.95) |  |
  Change from Week 7 to Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Change from Week 7 to Week 12 |  |  | -3.1 (2.13) | -4.7 (2.30)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.267, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = -1.3, 95% CI 2-sided [-3.5 to 1.0]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.609, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = -1.6, 95% CI 2-sided [-8.0 to 4.8]

6. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in NPI-C Rating Scale Subscale Scores for Disinhibition
Description: The NPI-C is used to rate the presence of neuropsychiatric symptoms across 12 domains. The 12 domains are collectively rated first by the informant/caregiver based on frequency (0-4), severity (0-3) & informant/caregiver distress (0-5), then by the participant based on frequency (0-4), which the clinician then integrates into a (0-3) clinical impression severity rating. The NPI-C disinhibition domain score is the sum of clinical impression severity scores for disinhibition questions 1-16, score ranges from 0-48, where higher score indicates greater clinical severity of symptom. LS mean was analyzed using MMRM analysis. Overall number analyzed=number of participants with data available for analysis. Number analyzed=number of participants with data available for analysis at the specified time point.
Time Frame: Stage 1: Baseline to Week 6; Stage 2: Week 7 to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 35 | 27 | 9 | 8
score on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 35 | 27 | 0 | 0
  Change from Baseline to Week 6 | -5.1 (0.82) | -5.4 (0.87) |  |
  Change from Week 7 to Week 12: number analyzed (Participants) | 0 | 0 | 9 | 8
  Change from Week 7 to Week 12 |  |  | -3.6 (1.35) | -2.4 (1.37)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.743, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = -0.3, 95% CI 2-sided [-2.4 to 1.7]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12: Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.575, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS Mean = 1.2, 95% CI 2-sided [-3.8 to 6.1]

7. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in Modified Clinical Global Impression of Severity (mCGI-S) Scale Scores
Description: mCGI-S is 7-point (1-7) scale requiring clinician to rate severity of participant's neurobehavioral disinhibition including aggression, agitation and irritability after NPI-C interview, at time of assessment relative to clinician's past experience with participants having same diagnosis. Considering total clinical experience, participant is assessed on severity of illness at time of rating as:0: not assessed;1: normal, not at all ill;2: borderline ill;3: mildly ill;4: moderately ill;5: markedly ill;6: severely ill;7: among most extremely ill participants. Higher score=increased severity. Negative change from baseline=improvement.LS mean was analyzed using analysis of covariance (ANCOVA) model. Overall number analyzed=participants with data available for analysis. Number analyzed=participants with data available for analysis at specified time point.
Time Frame: Stage 1: Baseline to Week 6; Stage 2: Week 7 to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 64 | 61 | 15 | 12
score on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 64 | 61 | 0 | 0
  Change from Baseline to Week 6 | -1.2 (0.16) | -1.3 (0.16) |  |
  Change from Week 7 to Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Change from Week 7 to Week 12 |  |  | -0.5 (0.36) | -1.1 (0.37)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6; Test type: Superiority; p = 0.664, ANCOVA; Difference in LS Mean = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12; Test type: Superiority; p = 0.273, ANCOVA; Difference in LS Mean = -0.6, 95% CI 2-sided [-1.9 to 0.6]

8. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in Patient Global Impression of Severity (PGI-S) Scores
Description: The PGI-S is a single-question scale used to assess the severity of symptoms of neurobehavioral disinhibition including aggression, agitation, and irritability, on a 7-point scale, as 1: normal, not at all ill; 2: borderline ill; 3: mildly ill; 4: moderately ill; 5: markedly ill; 6: severely ill; or 7: extremely ill. A higher score indicates worsening of the symptoms. Negative change from baseline indicates improvement. LS mean was analyzed using ANCOVA model. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Time Frame: Stage 1: Baseline to Week 6; Stage 2: Week 7 to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 62 | 61 | 15 | 12
score on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 62 | 61 | 0 | 0
  Change from Baseline to Week 6 | -1.1 (0.21) | -1.4 (0.20) |  |
  Change from Week 7 to Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Change from Week 7 to Week 12 |  |  | 0.0 (0.37) | -0.2 (0.41)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6; Test type: Superiority; p = 0.159, ANCOVA; Difference in LS Mean = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12; Test type: Superiority; p = 0.745, ANCOVA; Difference in LS Mean = -0.2, 95% CI 2-sided [-1.5 to 1.1]

9. Secondary Outcome: Stage 1 and Stage 2: Modified Clinical Global Impression of Change (mCGI-C) Raw Scores
Description: The mGCI-C is a scale that requires the clinician to rate the change of the participant's neurobehavioral disinhibition including aggression, agitation, and irritability at the time of assessment after the NPI-C interview, relative to the clinician's past experience with the participant's neurobehavioral disinhibition at admission. Considering total clinical experience, a participant is assessed for change of mental illness as: 0: not assessed; 1: very much improved; 2: much improved; 3: minimally improved; 4: no change; 5: minimally worse; 6: much worse; 7: very much worse. A higher score represents worsening of symptoms. Negative change from baseline indicates improvement.
Time Frame: Stage 1: Week 6; Stage 2: Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 63 | 61 | 15 | 12
score on a scale
  Week 6: number analyzed (Participants) | 63 | 61 | 0 | 0
  Week 6 | 2.7 (0.96) | 2.5 (0.91) |  |
  Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Week 12 |  |  | 3.0 (0.85) | 2.5 (1.17)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6; Test type: Superiority; p = 0.268, ANCOVA; Difference in LS Mean = -0.2, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12; Test type: Superiority; p = 0.147, ANCOVA; Difference in LS Mean = -0.5, 95% CI 2-sided [-1.2 to 0.2]

10. Secondary Outcome: Stage 1 and Stage 2: Patient Global Impression of Change (PGI-C) Raw Scores
Description: The PGI-C is a 7-point (1-7) scale used to assess treatment response, and it is rated as: 1: very much improved; 2: much improved; 3: minimally improved; 4: no change; 5: minimally worse; 6: much worse; 7: very much worse. A higher score indicates worsening of the symptoms. Negative change from baseline indicates improvement. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Time Frame: Stage 1: Week 6; Stage 2: Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: Placebo | Stage 1: AVP-786 | Stage 1: Placebo Non-responders to Stage 2: Placebo | Stage 1: Placebo Non-responders to Stage 2: AVP-786
Number analyzed (Participants) | 62 | 61 | 15 | 12
score on a scale
  Week 6: number analyzed (Participants) | 62 | 61 | 0 | 0
  Week 6 | 2.7 (1.17) | 2.4 (0.92) |  |
  Week 12: number analyzed (Participants) | 0 | 0 | 15 | 12
  Week 12 |  |  | 2.9 (1.03) | 2.6 (1.08)
Statistical Analysis 1: Comparison: Stage 1: Placebo vs Stage 1: AVP-786; Baseline to Week 6; Test type: Superiority; p = 0.655, ANCOVA; Difference in LS Mean = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 2: Comparison: Stage 1: Placebo Non-responders to Stage 2: Placebo vs Stage 1: Placebo Non-responders to Stage 2: AVP-786; Week 7 to Week 12; Test type: Superiority; p = 0.734, ANCOVA; Difference in LS Mean = -0.2, 95% CI 2-sided [-1.2 to 0.9]

ADVERSE EVENTS:
Time Frame: From start of study up to 7 days after the last dose of study drug (up to 13 weeks)
Description: Safety population- all participants who received at least one dose of study medication. As pre-specified in SAP, data was collected and reported by pooling the participants into one of the 2 arms based on the treatment received during the study (placebo / AVP-786). All Placebo arm includes participants who were treated with placebo in Stages 1, Stage 2, or both stages of the study. All AVP-786 arm includes participants who received AVP-786 throughout the study and only in Stage 2.
Groups:
- All Placebo: Participants received AVP-786 matching placebo capsules, orally, BID, during Stage 1 or Stage 2 of the study treatment.
- All AVP-786: Participants who were randomized to receive AVP-768 throughout the study and participants who were randomized to receive placebo in Stage 1 and were then re-randomized after Week 6 to receive AVP-786 in Stage 2.
  Participants received AVP-786-28/4.9 capsule along with AVP-786 matching placebo capsule, orally, QD for 1 week, followed by AVP-786-28/4.9 capsule, orally, BID, for the next one week and AVP-786-42.63/4.9 capsules (target dose), orally, BID during the rest of the treatment period.
Arm/Group | All Placebo | All AVP-786
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/83 | 3/115
Other Adverse Events (participants affected / at risk) | 4/83 | 7/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Placebo (N=83) | All AVP-786 (N=115)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Placebo (N=83) | All AVP-786 (N=115)
Dizziness (Nervous system disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03095066/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03095066/SAP_001.pdf